CLINICAL TRIAL: NCT04171089
Title: Suicide Prevention in Prepubertal Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 Pandemic
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Beth Brodsky, Associate Director, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7838
Record Dates: First submitted 2019-11-07; First posted 2019-11-20 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Suicidal Ideation; Suicide, Attempted
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted

STUDY DESIGN:
Intervention Model Description: Feasibility and acceptability of the Child Safety Planning Intervention among children and their parents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Child-Safety Plan Intervention (Experimental): A Child Safety Plan to prevent suicidal behavior will be developed with the children and their parents. The parents and child will complete feasibility and acceptability questionnaires.
  Interventions: Behavioral: Child- Safety Plan Intervention

INTERVENTIONS:
Behavioral: Child- Safety Plan Intervention — The intervention includes recognizing and knowing the individual's warning signs for a suicidal crisis, their personal coping/distraction skills, people to contact, as well as a restriction of the means to hurt oneself.

SUMMARY:
Suicidal ideation and behaviors are estimated to be as high as 4-16% and 1.5% (respectively) in the general 6-12-year-old population. However, there are currently no validated suicide prevention interventions specifically developed for this population.

This study aims to: (1) test the feasibility and acceptability of the Safety Planning Intervention for prepubertal Children (C-SPI) in 30 children (ages 6-12) who have made a suicide threat, suicidal behavior or reported suicidal ideation, and their parents, and (2) improve the investigator's understanding of suicidal ideation and behaviors in this age group. The results from the current project will be used to further develop the C-SPI, and to develop preliminary guidance and associated policy for clinicians to use.

DETAILED DESCRIPTION:
The Safety Planning Intervention (SPI) is a brief, protocol-driven and individually tailored tool that uses evidence-based practices for suicide prevention. The SPI aims to provide the individual with quick distraction and coping tools to overcome a suicidal crisis without acting upon the suicidal thoughts. The SPI was used in the Treatment for Adolescents Suicide Attempters study in youth 12-19 and has been found to be feasible and acceptable among adult patients and staff as well as among clinicians who work with adolescents. Its effectiveness in reducing suicide risk among veterans has also been confirmed. The SPI could be a good fit for children, as it uses concrete ways for the person to recognize their reaction, as well as concrete methods to cope with distress, which fits with the developmental stage of prepubertal children. Moreover, the collaborative way in which the personal safety plan is tailored to the suicidal person will allow the engagement of the child in the intervention. The SPI is an intervention that is relatively easy to administer and, therefore, if found to be appropriate for this age group, it could be implemented in different child-focused settings, including schools. The aim of the study is to evaluate the acceptability and feasibility of the Safety Planning Intervention for prepubertal Children's (C-SPI) among suicidal children and their parents. Additionally, children will be interviewed and be assessed for impulsivity, attention bias, irritability and coping skills.

ELIGIBILITY:
Inclusion Criteria:

* Suicidal thoughts or threats in the last six month or suicidal behavior in lifetime
* The child and his parent/guardian are English speakers
* Having a parent /guardian consent to the child participating in this study
* The clinician confirmed that the parents are suitable to take part in the intervention

Exclusion Criteria:

* Diagnosis of a psychotic disorder
* Intellectual disability

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Child-Safety Plan Intervention | Baseline
  The Patient Satisfaction Survey is a 12-item self-report questionnaire (child and parents versions), half of the items assess the feasibility of the child-safety plan intervention in this age group.
Acceptability of the Child-Safety Plan Intervention | Baseline
  The Patient Satisfaction Survey is a 12-item self-report questionnaire (child and parents versions), half of the items assess the acceptability of the child-safety plan intervention in this age group.

SECONDARY OUTCOMES:
Child's impulsivity | Baseline
  Child's impulsivity will be assessed using the "Go/No-go" computer task. The Go/No go is a measure of inhibitory control. An adaptation of the original Go/No go paradigm will be used, adjusted for elementary school children.
Child's symptoms of irritability | Baseline
  Child's symptoms of irritability will be assessed using the Affective Reactivity Index (ARI). The ARI is a seven-item scale that is both parent- and child-reported. The ARI asks about symptoms of irritability in the previous 6 months and includes an item assessing impairment due to irritability.
Child's attention bias | Baseline
  Child's attention bias will be evaluated using the Emotional picture dot prob computer task. The Emotional picture dot prob task is a spatially oriented, motivated attention task that capture the preattentive mechanism that automatically directs attention toward biologically relevant aversive stimuli, providing an indirect index of emotional reactivity.
Child's coping skills | Baseline
  Child's coping skills will be assessed using the Children's Response Styles Questionnaire. The Children's Response Styles Questionnaire consists of 25 items, each of which describes a particular response to symptoms of depression. For each item, children are asked to indicate how often they respond in this way when they are feeling sad. The items are grouped into two scales: (1) Ruminative Response subscale; and (2) Distracting Response subscale.
Child's conceptual level of death | Baseline
  Child's conceptual level of death will be assessed using the Death interview for children. The Death interview for children is an interview comprised of open-ended questions. It has been widely used to assess children's understanding of death as a biological event.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Stanley, PhD, Study Director — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brent DA, Greenhill LL, Compton S, Emslie G, Wells K, Walkup JT, Vitiello B, Bukstein O, Stanley B, Posner K, Kennard BD, Cwik MF, Wagner A, Coffey B, March JS, Riddle M, Goldstein T, Curry J, Barnett S, Capasso L, Zelazny J, Hughes J, Shen S, Gugga SS, Turner JB. The Treatment of Adolescent Suicide Attempters study (TASA): predictors of suicidal events in an open treatment trial. J Am Acad Child Adolesc Psychiatry. 2009 Oct;48(10):987-996. doi: 10.1097/CHI.0b013e3181b5dbe4. PMID 19730274
- [Result] Chesin MS, Stanley B, Haigh EA, Chaudhury SR, Pontoski K, Knox KL, Brown GK. Staff Views of an Emergency Department Intervention Using Safety Planning and Structured Follow-Up with Suicidal Veterans. Arch Suicide Res. 2017 Jan 2;21(1):127-137. doi: 10.1080/13811118.2016.1164642. Epub 2016 Apr 20. PMID 27096810
- [Result] Reyes-Portillo JA, McGlinchey EL, Toso-Salman J, Chin EM, Fisher PW, Mufson L. Clinician Experience and Attitudes Toward Safety Planning with Adolescents at Risk for Suicide. Arch Suicide Res. 2019 Apr-Jun;23(2):222-233. doi: 10.1080/13811118.2018.1456382. Epub 2019 Jan 12. PMID 29624113
- [Result] Stanley, B., & Brown, G. K. (2012). Safety planning intervention: a brief intervention to mitigate suicide risk. Cognitive and Behavioral Practice, 19(2), 256-264.
- [Result] Stanley B, Brown GK, Brenner LA, Galfalvy HC, Currier GW, Knox KL, Chaudhury SR, Bush AL, Green KL. Comparison of the Safety Planning Intervention With Follow-up vs Usual Care of Suicidal Patients Treated in the Emergency Department. JAMA Psychiatry. 2018 Sep 1;75(9):894-900. doi: 10.1001/jamapsychiatry.2018.1776. PMID 29998307
- [Result] Stanley B, Chaudhury SR, Chesin M, Pontoski K, Bush AM, Knox KL, Brown GK. An Emergency Department Intervention and Follow-Up to Reduce Suicide Risk in the VA: Acceptability and Effectiveness. Psychiatr Serv. 2016 Jun 1;67(6):680-3. doi: 10.1176/appi.ps.201500082. Epub 2016 Feb 1. PMID 26828397
- [Result] Stringaris A, Goodman R, Ferdinando S, Razdan V, Muhrer E, Leibenluft E, Brotman MA. The Affective Reactivity Index: a concise irritability scale for clinical and research settings. J Child Psychol Psychiatry. 2012 Nov;53(11):1109-17. doi: 10.1111/j.1469-7610.2012.02561.x. Epub 2012 May 10. PMID 22574736
- [Result] Kimonis ER, Frick PJ, Fazekas H, Loney BR. Psychopathy, aggression, and the processing of emotional stimuli in non-referred girls and boys. Behav Sci Law. 2006;24(1):21-37. doi: 10.1002/bsl.668. PMID 16491477
- [Result] Abela, J. R. Z., Rochon, A., & Vanderbilt, E. (2000). The Children's Response Style Questionnaire (Unpublished questionnaire). Montreal, Canada: McGill University